CLINICAL TRIAL: NCT05839041
Title: A Single and Multiple Dose Study to Evaluate Safety, Pharmacokinetics, and Treatment Effect of Intravitreal AVD-104 in Participants With Geographic Atrophy Secondary to Age-related Macular Degeneration
Brief Title: A Multiple Dose Study of AVD-104 for Geographic Atrophy (GA) Secondary to Age-Related Macular Degeneration (AMD)
Acronym: SIGLEC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Aviceda Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVD-104-C01
Record Dates: First submitted 2023-04-10; First posted 2023-05-03 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-11

CONDITIONS: Geographic Atrophy of the Macula; Macular Degeneration
Keywords: Age-related Macular Degeneration; Geographic Atrophy; Dry AMD
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Intervention Model Description: Part 1 - Open Label, Multi-Center, Dose Escalation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part 2 - Double Masked, Randomized, Multi-Center
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part 1 (Experimental): Participants will receive a single intravitreal injection of AVD-104 at one of 4 escalating doses. All participants will be followed up for safety until Month 3.
  Interventions: Drug: AVD-104
- Part 2: High dose AVD-104 (Active Comparator): 100 participants will be randomized and treated with bimonthly intravitreal injections of high-dose AVD-104 for the first 12 months. They will continue bimonthly injections for months 13-24.
  Interventions: Drug: AVD-104
- Part 2: Low dose AVD-104 (Active Comparator): 100 participants will be randomized and treated with monthly intravitreal injections of low dose AVD-104 for 24 months.
  Interventions: Drug: AVD-104
- Part 2: Avacincaptad (Active Comparator): 100 participants will be randomized to receive monthly injections of avacincaptad (2 mg. intravitreal)
  Interventions: Drug: Avacincaptad

INTERVENTIONS:
Drug: AVD-104 — Intravitreal injection
  Arms: Part 1; Part 2: High dose AVD-104; Part 2: Low dose AVD-104
Drug: Avacincaptad — Intravitreal injection of 2 mg avacincaptad
  Arms: Part 2: Avacincaptad

SUMMARY:
Investigate the Safety, Pharmacokinetics, and Treatment effects of Single and Multi-dose of Intravitreal AVD-104 in participants with geographic atrophy secondary to age-related macular degeneration.

DETAILED DESCRIPTION:
Part 1 of the trial will be a multi-center, open label safety and dose escalation study with a potential enrollment of 30 participants having geographic atrophy (GA) secondary to macular degeneration. They will receive a single intravitreal injection of study drug (AVD-104) and will be followed for 3 months for safety observation. They will have both aqueous humor and peripheral blood drawn for pharmacokinetic and pharmacodynamic evaluations.

Part 2 will be a multi-center, double masked, randomized trial to evaluate the treatment effect of AVD-104 on participants with geographic atrophy secondary to macular degeneration. Participants will be randomized to high dose AVD-104, low dose AVD-104, or active comparator (avacincaptad). The primary endpoint will be the difference in the rate of growth of the GA area as measured by fundus autofluorescence.

ELIGIBILITY:
Inclusion Criteria:

Part 1:

1. BCVA in the study eye using ETDRS Chart Visual Acuity Scale (VAS) of 5 to 55 letters (equivalent to Snellen VA of approximately 20/800 - 20/80)
2. If GA is multifocal, at least one focal lesion must be ≥ 1.25 mm2 (0.5 DA)
3. GA may be center involved.

Part 2:

1. BCVA in the study eye using ETDRS Chart VAS of 24 letters or better (equivalent to Snellen VA of 20/320 or better)
2. Confirmed diagnosis of AMD that is non-center involving (i.e., non-sub-foveal) GA in 50% of participants. Center involvement allowed in 50% of participants.
3. The entire GA lesion must be completely visualized on the macula centered image and must be able to be imaged in its entirety and not contiguous with any areas of peripapillary atrophy.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Part 1 and 2

- Presence of the following ocular conditions - in the Study Eye:

1. Exudative AMD or choroidal neovascularization (CNV), including any evidence of retinal pigment epithelium rips or evidence of neovascularization anywhere based on spectral domain optical coherence tomography (SD-OCT) imaging and/or fluorescein angiography as assessed by the Reading Center.
2. Any ocular condition other than GA secondary to AMD that may require surgery or medical intervention during the study period or, in the opinion of the Investigator, could compromise visual function during the study period.

Ages: 55 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Dose Limiting Toxicity in Part 1 | 3 months
  The number of participants experiencing a dose limiting toxicity corresponding to a category of 3 or greater on the National Cancer Institute Common Terminology Criteria for Adverse Events
The Rate of Change in Area of Geographic Atrophy at Month 12 in Participants in Part 2 | 12 months
  The rate of change from baseline in area of GA as measured by fundus autofluorescence at month 12.

SECONDARY OUTCOMES:
Prevention of Vision Loss from Baseline in Participants in Part 2 | 12 months
  Proportion of participants with 15 or greater letter loss in best corrected visual acuity (BCVA) (assessed with the Early Treatment Diabetic Retinopathy Study [ETDRS] visual acuity).

CONTACTS AND LOCATIONS:
Overall Officials: David Callanan, MD, Study Director — Aviceda Therapeutics
Locations (55):
- United States (55):
  - Associated Retina Consultants, Gilbert, Arizona
  - Arizona Retina and Vitreous Consultants, Phoenix, Arizona
  - Associated Retina Consultants, Scottsdale, Arizona
  - Retina Vitreous Associates Medical Group, Beverly Hills, California
  - Macula & Retina Institute, Glendale, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - Kaiser Permanente, Riverside, California
  - Retinal Consultants Medical Group, Inc., Sacramento, California
  - Retinal Consultants Medical Group, Sacramento, California
  - West Coast Retina, San Francisco, California
  - RCA: California Retina Consultants, Santa Barbara, California
  - Retina Group of New England, PC, Waterford, Connecticut
  - Rand Eye Institute, Deerfield Beach, Florida
  - Retina Group of Florida, Fort Lauderdale, Florida
  - Florida Retina Institute, Orlando, Florida
  - Retina Specialty Institute, Pensacola, Florida
  - Retina Vitreous Associates of Florida, St. Petersburg, Florida
  - Southern Vitreoretinal Associates, Tallahassee, Florida
  - Center for Retina & Macular Disease, Winter Haven, Florida
  - Southeast Retina Center, Augusta, Georgia
  - University Retina and Macula Associates, Chicago, Illinois
  - Illinois Retina Associates, Oak Park, Illinois
  - Midwest Eye Institute, Indianapolis, Indiana
  - Cumberland Valley Retina Consultants, Hagerstown, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - New England Retina Consultants, Springfield, Massachusetts
  - Retina Specialists of Michigan, Grand Rapids, Michigan
  - Associated Retinal Consultants, Royal Oak, Michigan
  - Retina Consultants of Minnesota, Minneapolis, Minnesota
  - Mississippi Retina Associates, Jackson, Mississippi
  - Sierra Eye Associates, Reno, Nevada
  - Retina Center of New Jersey, Bloomfield, New Jersey
  - NJ Retina, Edison, New Jersey
  - Retina-Vitreous Surgeons of Central NY, Syracuse, New York
  - Long Island Vitreoretinal Consultants, Westbury, New York
  - North Carolina Retina Associates, Wake Forest, North Carolina
  - Retina Associates of Cleveland, Inc, Beachwood, Ohio
  - Retina Associates of Cleveland, Cleveland, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Mid-Atlantic Retina, Bethlehem, Pennsylvania
  - Erie Retina Research, LLC, Erie, Pennsylvania
  - Retina Consultants of Charleston, Charleston, South Carolina
  - Palmetto Retina Center, West Columbia, South Carolina
  - Tennessee Retina, Nashville, Tennessee
  - Retina Research Institute of Texas Abilene TX, Abilene, Texas
  - Texas Retina Associates, Arlington, Texas
  - Austin Retina Associates, Austin, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Texas Retina Associates, Dallas, Texas
  - Texas Retina Associates, Fort Worth, Texas
  - Valley Retina Institute, McAllen, Texas
  - Retina Consultants of Texas, San Antonio, Texas
  - Retina Consultants of Texas, The Woodlands, Texas
  - Rocky Mountain Retina Consultants, Salt Lake City, Utah
  - Spokane Eye Clinic, Spokane, Washington